CLINICAL TRIAL: NCT04284956
Title: Major Leg Wound Complications Between the Proximal and Distal Segments of Saphenous Veins Harvested by No-Touch Technique in Coronary Artery Bypass Graft Surgery: a Single-center Randomized Within-subject Controlled Clinical Trial
Brief Title: Proximal Versus Distal Segments of No-Touch Saphenous Vein Grafts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-F06
Record Dates: First submitted 2020-02-22; First posted 2020-02-26 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Leg Wound Complication After No-Touch Harvestingof Veins
Keywords: leg wound complication; No-Touch saphenous vein harvesting technique; coronary artery bypass graft

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proximal group (Experimental): Proximal segment of saphenous veins are harvested from the thigh by No-Touch technique and randomized to bypass the left or right territory of coronary system
  Interventions: Procedure: Proximal and distal segment of saphenous vein harvested by No-Touch technique
- Distal group (Active Comparator): Distal segment of saphenous veins are harvested from the shank of the ipsilateral leg by No-Touch technique and used to bypass the right or left territory of coronary system (depending on the randomizing result of the proximal segments)
  Interventions: Procedure: Proximal and distal segment of saphenous vein harvested by No-Touch technique

INTERVENTIONS:
Procedure: Proximal and distal segment of saphenous vein harvested by No-Touch technique — two longitudinal incisions are made on the thigh and shank from unilateral lower limb (for harvesting of proximal segment of saphenous vein, incision is started from about 3 or 4cms inferolateral to the pubic tubercle and then extended downward). As previous reported. the adventitia and perivascular tissue are carefully kept intact to avoid damage. Then a margin of about 5 mm from both sides of the vein is created to include the fat pedicle using electrocautery, and all visible side branches are ligated with 4-0 silk or by metal clipping (branches are divided at the pedicle margin rather than the vein trunk). The saphenous vein is then separated from its bed using scissors and electrocautery, together with surrounding tissue.

SUMMARY:
The optimum segment of No-Touch veins for bypassing is still undefined. The purpose of this study is to assess the incidence of leg wound complication after No-Touch harvesting of proximal segment of saphenous veins compared to distal segment of veins in the leg. Graft occlusion rates between the two segments of veins for bypassing will also be compared during follow-up.

DETAILED DESCRIPTION:
This is a prospective, single-center, open-label, randomized within-subject-controlled trial. We aim to randomize 100 patients undergoing isolated coronary artery bypass graft (CABG). We consecutively screen patients during the study enrollment period and seek informed consent from all eligible patients. In each patient, one saphenous vein graft (SVG) will be randomized to be the proximal segment, while another will be the distal segment as control. Healing of leg wounds will be assessed on day 6 post-operatively. Follow-up will be performed via face-to-face interview until at least 1 year after the operation by CT angiography.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older who undergo primary isolated open-chest CABG with two vein grafts, one to the left coronary territory and the other to the right, with or without cardiopulmonary bypass

Exclusion Criteria:

* Concomitant cardiac or vascular surgeries (i.e. valve repair or replacement, Maze surgery)
* Redo CABG
* Emergent CABG (cardiogenic shock, inotropic pressure support, IABP)
* Severe vein varicosity as assessed after vein harvesting and before randomization
* Use of vascular stapler for anastomosis
* Endarterectomy of coronary artery during surgery
* Left ventricular repair due to ventricular aneurysm
* Concomitant life-threatening disease likely to limit life expectancy to less than two years
* Severe renal insufficiency (i.e. creatinine >200 μmol/L)
* Contraindications for dual antiplatelet therapy, such as active gastroduodenal ulcer
* Participant of other ongoing clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Major leg wound complication at 6 days postoperatively | 6 days postoperatively
  a leg wound that had failed to respond to conservative treatment and required subsequent surgical intervention such as debridement, re-suture, delayed wound closure

SECONDARY OUTCOMES:
Major leg wound complication during 3-month follow-up | 3 month
  a leg wound that had failed to respond to conservative treatment and required subsequent surgical intervention such as debridement, re-suture, delayed wound closure
Graft vessel occlusion at 3 month and 1 year | 3 months and 1 year
  Graft occlusion is detected by multislice computed tomography angiography (MSCTA). Graft assessment is conducted according to the FitzGibbon criteria. Each graft is graded as A (excellent), B (fair), or O (occluded). Contrast filling of the grafts, anastomoses, and coronary arteries beyond the graft are considered in each assessment. Grade A indicates that the graft is patent with ≤50% stenosis. Grade B indicates that graft stenosis is >50% but not occluded. When a conduit does not fill with contrast at all, it is considered Grade O and included with string sign found in any segment (including proximal anastomotic site, distal anastomotic site, and main trunk). Both of these latter findings are considered together and referred to as occlusion in the analysis.

OTHER OUTCOMES:
Major adverse cardiac or cerebrovascular events (MACCE) | 3 months and 1 year
  including cardiovascular death, non-fatal myocardial infarction (MI), stroke and target vessel revascularization
Individual MACCE | 3 months and 1 year
  including cardiovascular death, non-fatal myocardial infarction, stroke and target vessel revascularization
Recurrence of angina | 3 months and 1 year
  Events that fulfill the following definition are to be coded as Angina:
  i. ischemic chest pain or equivalent (e.g. arm, neck or jaw pain or discomfort thought to be related to cardiac ischemia); and ii. no evidence of MI; and iii. no clear alternative (non-cardiac) explanation (e.g. anemia, arrhythmia)

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital Chinese Academay of Medical Science and National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No